CLINICAL TRIAL: NCT06794541
Title: Multicenter, Open-label Trial to Evaluate the Safety and Tolerability of Intravenous Eravacycline in Pediatric Patients From 8 Years to Less Than 18 Years of Age With Complicated Intra-abdominal Infections (cIAI)
Brief Title: A Study to Evaluate the Safety and Tolerability of Eravacycline in Pediatric Patients Aged 8 to 17 With Complicated Intra-abdominal Infections (cIAI)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tetraphase Pharmaceuticals, Inc (Industry)
Collaborators: Innoviva Specialty Therapeutics (Industry)
Responsible Party: Sponsor
Organization: Innoviva Specialty Therapeutics (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS434-2023-001
Record Dates: First submitted 2025-01-15; First posted 2025-01-27 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Complicated Intra-abdominal Infections (cIAI)
Keywords: Complicated Intra-abdominal Infections; cIAI; eravacycline
MeSH Terms: interventions — eravacycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: Cohort 1 (Experimental): Eravacycline intravenous formulation will be administered as a single 60-minute IV infusion for participants 12 to <18 years of age
  Interventions: Drug: Eravacycline 1.5mg/kg
- Experimental: Cohort 2a (Experimental): Eravacycline intravenous formulation will be administered as a single 60-minute IV infusion for participants 10 to <12 years of age
  Interventions: Drug: Eravacycline 2mg/kg
- Experimental: Cohort 2b (Experimental): Eravacycline intravenous formulation will be administered as a single 60-minute IV infusion for participants aged 8 to <10 years of age
  Interventions: Drug: Eravacycline 2mg/kg

INTERVENTIONS:
Drug: Eravacycline 2mg/kg — intravenous (IV) infusion
  Arms: Experimental: Cohort 2a; Experimental: Cohort 2b
Drug: Eravacycline 1.5mg/kg — intravenous (IV) infusion
  Arms: Experimental: Cohort 1

SUMMARY:
A Phase 2 trial to assess safety, tolerability, and pharmacokinetics of eravacycline in pediatric patients aged 8 to <18 years with cIAI.

ELIGIBILITY:
Inclusion Criteria:

1. Children from 8 to <18 years of age (as of the day of the informed consent [and assent, if applicable] is obtained), hospitalized for cIAI with one of the following diagnoses:

   1. Intra-abdominal abscess (including hepatic and splenic abscesses).
   2. Gastric or intestinal perforation associated with diffuse peritonitis.
   3. Peritonitis: diffuse infection of the peritoneum (but not spontaneous bacterial peritonitis associated with cirrhosis and chronic ascites).
   4. Appendicitis with perforation, peritonitis, or abscess (complicated appendicitis).
   5. Cholecystitis with perforation or abscess.
2. Patient has evidence of age-appropriate abnormal systemic inflammatory response syndrome
3. Written informed consent from parent(s) or other legally authorized representative(s) and assent (according to local requirements).
4. In the investigator's opinion, the patient will require hospitalization for at least 4 days.
5. The patient must require hospitalization initially and antibacterial therapy for 4 to 14 days in addition to surgical intervention for the treatment of the current cIAI based on the judgment of the investigator.
6. The patient has sufficient intravascular access (peripheral or central) to receive eravacycline.
7. The patient meets either (A or B) of the following criteria:

   1. Pre-operative enrollment:

      * i. Has a sonogram or radiographic imaging result consistent with the diagnosis of cIAI, and
      * ii. Acute surgical or percutaneous intervention (open laparotomy, laparoscopic surgery, or percutaneous drainage of an abscess) is foreseen within 24 hours.

      OR
   2. Intra-operative/postoperative enrollment:

      * i. Visual confirmation of cIAI (presence of pus within the abdominal cavity), and
      * ii. Surgical intervention includes open laparotomy, laparoscopic surgery, or percutaneous draining of an abscess, and
      * iii. Intervention is considered adequate by the surgical team.

Exclusion Criteria:

1. Patient is considered by the investigator to be unlikely to survive the trial period, and/or has any rapidly progressing disease or immediately life-threatening illness.
2. Patient's laboratory test results reveal alanine aminotransferase or aspartate transaminase >5×upper limit of normal range (ULN).
3. Patient's laboratory test results reveal total bilirubin >2×ULN, unless isolated hyperbilirubinemia is directly related to the acute process.
4. Patient requires peritoneal dialysis, hemodialysis, or hemofiltration at screening. Patient has an estimated glomerular filtration rate (eGFR) <50 mL/minute/1.73 m².
5. Patient has previously received eravacycline or have enrolled previously in the current trial and been discontinued.
6. Patient has evidence or history of a clinically significant medical condition that may, in the opinion of the investigator, impair trial participation or pose a significant safety risk or diminish the patient's availability to undergo all trial procedures and assessments.
7. Patient is likely to require more than 14 days of treatment with eravacycline, in the opinion of the investigator.
8. Patient is currently participating in or has participated in an interventional clinical trial with an investigational compound or device within 30 days or <5 half-lives of the eravacycline (whichever is longer) prior to screening.
9. Patient has immunocompromised condition, including acquired immune deficiency syndrome (AIDS), organ (including bone marrow) transplant recipients, and hematologic malignancy, or receiving immunosuppressive therapy, including cancer chemotherapy, medications for prevention of organ transplantation rejection, or chronic administration of systemic corticosteroids (defined as the systemic equivalent of ≥2 mg/kg total daily dose of prednisone for patients ≤20 kg, or >40 mg of prednisone per day for patients >20 kg, administered continuously for more than 14 days in the 30 days prior to the first dose of eravacycline.
10. Patient has known or suspected inflammatory bowel disease.
11. Patient has pancreatitis.
12. Patient has systemic malignancy that required chemotherapy, immunotherapy, radiation therapy, or antineoplastic therapy within the previous 3 months.
13. Patient has history of hypersensitivity or allergic reaction to any tetracycline antibiotics.
14. Patient has cIAI caused by a pathogen(s) resistant to eravacycline at screening.
15. Patient has received antibacterial drug therapy for continuous duration of >72 hours immediately preceding screening unless they are considered treatment failures. Note: Treatment failure is defined as persistent fever and/or clinical symptoms or the development of a new intra-abdominal abscess after ≥72 hours of antibiotic therapy.
16. Patient has received any tetracycline within 14 days of screening.
17. Patient used cytochrome P450 (CYP) 3A inducers or inhibitors within 14 days of screening or is receiving or anticipated to need treatment with CYP3A inducers or inhibitors during the treatment period.
18. Patient used inducers and/or inhibitors of P-glycoprotein (P-gp), organic anion transporting polypeptide (OATP)1B1, and OATP1B3 transporters within 14 days of screening or is receiving or anticipated to need treatment such agents during the treatment period.
19. Patient is currently using or anticipates use of anticoagulant therapy during the treatment period.
20. Patient is unable or unwilling, in the opinion of the investigator, to comply with the protocol.
21. Patients who are known to be pregnant (positive pregnancy test) and/or breastfeeding at the time of screening.
22. Sexually active patients of childbearing potential (those with menarche and/or thelarche) who are unwilling or unable to use an acceptable method of contraception (at least 2 medically accepted, effective methods of birth control [e.g., condom, oral contraceptive, indwelling intrauterine device, hormonal implant/patch, injections, approved cervical ring]) or sexual abstinence.
23. Patient has any other circumstance that, in the opinion of the investigator, precludes the patient's participation in the trial.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Estimated)
Dates: Start 2025-05-22 (Actual); Primary Completion 2029-02-17 (Estimated); Study Completion 2029-03-19 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with Adverse Events (AEs) from the first dose of any amount of eravacycline | 28 days
Change from baseline values over time in electrocardiogram (ECG) QT measurements | Day 28
Change from baseline values over time in diastolic blood pressure | Day 28
Change from baseline values over time in systolic blood pressure | Day 28
Change from baseline values over time in liver function tests assessed by Comprehensive Metabolic Panel (CMP) | Day 28
Change from baseline values over time of hemoglobin | Day 28
Change from baseline values over time in white blood count | Day 28
Change from baseline values over time in platelets | Day 28
Change from baseline values over time in kidney function assessed by CMP | Day 28

SECONDARY OUTCOMES:
Steady state area under the curve (AUC (0-24)) of eravacycline | Dose cycle 4 (each dose cycle is 24 hours)
Steady state maximum concentration (Cmax) of eravacycline | Dose cycle 4 (each dose cycle is 24 hours)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - UCLA Ronald Reagan University of California Los Angeles Medical Center, Los Angeles, California
  - Children's Hospital of Orange County, Orange, California
  - Ann and Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Children's Hospital of LSU Health Sciences Center Shreveport, Shreveport, Louisiana
  - West Virginia University Medicine Children's Hospital, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests may be submitted starting 6 months after primary article publication and the data will be made accessible for up to 24 months; extensions may be considered on a case-by-case basis
Access Criteria: Subject to certain criteria, conditions, and exceptions and upon completion of the review and approval of the Research Proposal and Statistical Analysis Plan, Qualified Researchers engaging in independent scientific research can be provided de-identified IPD following the execution of a Data Sharing Agreement